CLINICAL TRIAL: NCT05936749
Title: Pre-implantation Genetic Testing for Monogenic Disease: Single Center Experience
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 14/23
Record Dates: First submitted 2023-06-14; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Genetic Disease; Aneuploidy
MeSH Terms: conditions — Genetic Diseases, Inborn; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Pre-implantation genetic testing

SUMMARY:
This monocentric retrospective observational study aims to evaluate the efficacy of pre-implantation genetic testing for monogenic diseases (PGT-M). The effectiveness will be assessed in terms of live birth rate (LBR), cumulative live birth rate (CLBR) per couple, and abortion rate (AR). Considering how many cycles the participants have undergone to achieve a viable blastocyst. The secondary objective is to evaluate the incidence of aneuploidy in unaffected embryos, in order to understand the need for pre-implantation genetic testing for aneuploidy (PGT-A)in addition to PGT-M.

ELIGIBILITY:
Inclusion Criteria:

* Patients fertile or infertile that have undergone preimplantation genetic testing for monogenic diseases (PGTM).

Exclusion Criteria:

* No exclusion criteria will be taken into consideration.

Ages: 34 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: All 76 participants that underwent PGTM testing in the Fertility Center starting from the beginning of 2016 all through the end of 2022, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Live birth rate (LBR) | 7 years of inclusion
  LBR will be measured as a percentage
Cumulative live birth rate (CLBR) per couple | 7 years of inclusion
  CLBR per couple will be measured as a percentage
Abortion rate (AR) | 7 years of inclusion
  AR will be measured as a percentage

SECONDARY OUTCOMES:
Aneuploidy | 7 years of inclusion
  Aneuploidy embryo rate will be measured as a percentage

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT05936749/Prot_000.pdf
  • Informed Consent Form (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT05936749/ICF_001.pdf